CLINICAL TRIAL: NCT05066295
Title: Strengthening Families to Prevent Child Neglect and Abuse With Community Based Protective Approaches: Culturally Appropriate Program Development and Educational Design
Brief Title: Validation and Reliability of the Parents Assessment of Protective Factors Survey
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Perran Boran, Professor of Pediatrics, Marmara University
Other Study IDs: 09.2021.848
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Family
Keywords: parents' assessment; protective factors; child abuse; prevention; validity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neglect and abuse, which have a devastating effect on children, can be prevented with community-based education programs aimed at strengthening families. The study aimed to validate and determine reliability of the "Parents Assessment of Protective Factors (PAPF) survey" and to develop a culturally appropriate program and educational design for strengthening families.

DETAILED DESCRIPTION:
The American Center for Social Policy Studies (CSSP) Center for Quality Improvement in Early Childhood (QIC_EC) defined protective factors that will form the basis of programs designed to prevent neglect and abuse, with community-based approaches. Community-based programs for primary prevention should be developed to prevent neglect and abuse, before it occurs. Existing studies in our country show that there is rarely a focus on preventing adverse childhood experiences with primary preventive approaches. Most of the studies are school-based, and aimed at increasing awareness of children and families about abuse.

This study aimed to evaluate the Turkish translation of the PAPF survey for validity and reliability and to adapt a culturally appropriate program and educational design for strengthening families, with a multidisciplinary team.

In the first step of the study, Turkish validity and reliability of the Parents Assessment of Protective Factors (PAPF) survey, will be conducted and applied to parents to determinate the protective factors. Turkish version of Adverse Childhood Experience Questionnaire (ACE), will be applied simultaneously with the PAPF survey, to identify adverse childhood experiences of parents that might affect parental resilience, parenting characteristics, and family dynamics.

In the second phase of the study, community-based family education programs that are currently being implemented in different countries will be reviewed by a multidisciplinary team (healthcare professionals, social workers and non-governmental organizations). A culturally appropriate educational primary prevention program for child neglect and abuse will be developed.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children aged between 0 to 8 years
* Ability to read and complete the self-assessment questionnaires

Exclusion Criteria:

* Parents who do not give consent to participate in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Parents of children aged between 0 to 8 years
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Turkish Validation of The Parents Assessment of Protective Factors (PAPF) Survey | Baseline
  Parents Assessment of Protective Factors (PAPF) Survey will be validated
Turkish Reliability of The Parents Assessment of Protective Factors (PAPF) Survey | Baseline
  Parents Assessment of Protective Factors (PAPF) Survey will be tested for reliability
Turkish Reliability of The Parents Assessment of Protective Factors (PAPF) Survey | at 6 months
  Parents Assessment of Protective Factors (PAPF) Survey will be tested for reliability

SECONDARY OUTCOMES:
Subscale scores for each protective factors | Baseline
  Parents Assessment of Protective Factors (PAPF) Survey subscale scores will be computed. Higher scores indicate greater protective factors.
Protective Factors Index (PFI) | Baseline
  Parents Assessment of Protective Factors (PAPF) Survey total scores will be summed
Adverse Childhood Events | Baseline
  Adverse Childhood Events will be measured with Adverse Childhood Events Questionnaire.
  Higher scores indicate increased exposure to trauma, which have been associated with a greater risk of negative consequences.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Requests for wider sharing of data (for example in response to publications about the study and willingness to share), will be addressed on a case-by-case basis. Any data sharing request will be made to investigators through a pre-defined data requisition form. This form will contain information about the applicant, institution, purpose of data request, study objectives, ethical clearance of the study, etc. Once a request has been made the data governance body will discuss if that request was appropriate; data will be released following signing of the data sharing agreement. The data will be stored on the Marmara University servers and not be deposited in any 'community' database.